CLINICAL TRIAL: NCT04977336
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Dose-ranging, Study Evaluating the Efficacy and Safety of VX-548 for Acute Pain After a Bunionectomy
Brief Title: A Study Evaluating Efficacy and Safety of VX-548 for Acute Pain After a Bunionectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX21-548-101
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Participants received placebo matched to VX-548 and Hydrocodone bitartrate/acetaminophen (HB/APAP) for 2 days.
  Interventions: Drug: Placebo (matched to VX-548); Drug: Placebo (matched to HB/APAP)
- HB/APAP (Active Comparator): Participants received HB 5 milligrams (mg)/ APAP 325 mg every 6 hours (q6h) for 2 days.
  Interventions: Drug: HB/APAP
- VX-548: Low Dose (Experimental): Participants received VX-548 20 mg as first dose, followed by VX-548 10 mg tablet every 12 hours (q12h) for 2 days.
  Interventions: Drug: VX-548
- VX-548: Mid Dose (Experimental): Participants received VX-548 60 mg as first dose, followed by VX-548 30 mg q12h for 2 days.
  Interventions: Drug: VX-548
- VX-548: High Dose (Experimental): Participants received VX-548 100 mg as first dose, followed by VX-548 50 mg q12h for 2 days.
  Interventions: Drug: VX-548

INTERVENTIONS:
Drug: VX-548 — Tablets for oral administration.
  Other Names: Suzetrigine
  Arms: VX-548: High Dose; VX-548: Low Dose; VX-548: Mid Dose
Drug: HB/APAP — Capsules for oral administration.
  Arms: HB/APAP
Drug: Placebo (matched to VX-548) — Placebo matched to VX-548 for oral administration.
  Arms: Placebo
Drug: Placebo (matched to HB/APAP) — Placebo matched to HB/APAP for oral administration.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of VX-548 doses in treating acute pain after a bunionectomy.

ELIGIBILITY:
Key Inclusion Criteria:

* Before Surgery:

  * Participant scheduled to undergo a primary unilateral bunionectomy with distal first metatarsal osteotomy (i.e., Austin procedure) and internal fixation under regional anesthesia (Mayo and popliteal sciatic block)
* After Surgery:

  * Participant is lucid and able to follow commands
  * All analgesic guidelines were followed during and after the bunionectomy

Key Exclusion Criteria:

* Before Surgery:

  * Prior history of bunionectomy or other foot surgery on the index foot
  * History of cardiac dysrhythmias requiring anti-arrhythmia treatment(s)
  * Any prior surgery within 1 month before the first study drug
* After Surgery:

  * Participant had a Type 3 deformity requiring a base wedge osteotomy or concomitant surgery such as hammertoe repair, or had medical complications during the bunionectomy that, in the opinion of the investigator, should preclude randomization

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Shoals Medical Trials Inc., Sheffield, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Anaheim Clinical Trials, Anaheim, California
  - Lotus Clinical Research, Pasadena, California
  - New Hope Research Development, Tarzana, California
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Chesapeake Research Group, Pasadena, Maryland
  - Midwest Clinical Research Center, Dayton, Ohio
  - First Surgical Hospital, Bellaire, Texas
  - Legent Orthopedic Hospital, Carrollton, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - JBR Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

REFERENCES:
- [Derived] Jones J, Correll DJ, Lechner SM, Jazic I, Miao X, Shaw D, Simard C, Osteen JD, Hare B, Beaton A, Bertoch T, Buvanendran A, Habib AS, Pizzi LJ, Pollak RA, Weiner SG, Bozic C, Negulescu P, White PF; VX21-548-101 and VX21-548-102 Trial Groups. Selective Inhibition of NaV1.8 with VX-548 for Acute Pain. N Engl J Med. 2023 Aug 3;389(5):393-405. doi: 10.1056/NEJMoa2209870. PMID 37530822
- [Derived] Russo MA, Baron R, Dickenson AH, Kern KU, Santarelli DM. Ambroxol for neuropathic pain: hiding in plain sight? Pain. 2023 Jan 1;164(1):3-13. doi: 10.1097/j.pain.0000000000002693. Epub 2022 May 17. PMID 35580314

RESULTS

PARTICIPANT FLOW:
Groups:
- VX-548: Low Dose: Participants received VX-548 20 mg as first dose, followed by VX-548 10 mg every 12 hours (q12h) for 2 days.
Period: Overall Study
Arm/Group | Placebo | HB/APAP | VX-548: Low Dose | VX-548: Mid Dose | VX-548: High Dose
Started | 59 | 60 | 33 | 62 | 60
Completed | 58 | 60 | 32 | 61 | 58
Not Completed | 1 | 0 | 1 | 1 | 2
Not completed — Withdrawal of Consent (not due to AE) | 1 | 0 | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug.
Groups:
- Placebo: Participants received placebo matched to VX-548 and HB/APAP for 2 days.
- HB/APAP: Participants received HB 5 mg/ APAP 325 mg q6h for 2 days.
- VX-548: Low Dose: Participants received VX-548 20 mg as first dose, followed by VX-548 10 mg q12h for 2 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | HB/APAP | VX-548: Low Dose | VX-548: Mid Dose | VX-548: High Dose | Total
Number analyzed (Participants) | 59 | 60 | 33 | 62 | 60 | 274
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (13.6) | 50.0 (12.5) | 47.8 (15.5) | 48.3 (13.1) | 47.6 (13.7) | 48.4 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 50 | 25 | 57 | 53 | 234
  Male | 10 | 10 | 8 | 5 | 7 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 22 | 6 | 20 | 21 | 86
  Not Hispanic or Latino | 42 | 38 | 27 | 42 | 39 | 188
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 2 | 3
  Asian | 3 | 3 | 2 | 0 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 13 | 13 | 9 | 17 | 14 | 66
  White | 41 | 44 | 22 | 44 | 42 | 193
  More than one race | 1 | 0 | 0 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Pain Intensity at Baseline (at 0 hours) as Recorded on Numeric Pain Rating Scale (NPRS) [Mean (Standard Deviation); unit: units on a scale] — Pain intensity was recorded on 11-point NPRS, score range: 0 to 10, where 0=no pain and 10=worst imaginable pain.
  units on a scale | 6.9 (1.7) | 6.9 (1.9) | 6.9 (1.8) | 6.6 (1.8) | 6.7 (1.7) | 6.8 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Time-Weighted Sum of Pain Intensity Difference (SPID) as Recorded on a Numeric Pain Rating Scale (NPRS) 0 to 48 Hours (SPID48) After the First Dose of Study Drug
Description: SPID was calculated as the sum of the product of time (in hours) elapsed since previous measurements and pain intensity difference. Pain intensity difference was calculated by subtracting the pain intensity score at given post-dose time points from the baseline pain intensity scores (using pain rating score range: 0= no pain to 10= worst possible pain). SPID48 was calculated from 0 to 48 hours and the score range was -480 (worst score) to 480 (best score).
Time Frame: 0 to 48 hours After First Dose of Study Drug
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- HB/APAP: Participants received HB 5 mg/ APAP 325 mg every q6h for 2 days.
Arm/Group | Placebo | HB/APAP | VX-548: Low Dose | VX-548: Mid Dose | VX-548: High Dose
Number analyzed (Participants) | 59 | 60 | 33 | 62 | 60
units on a scale | 100.98 (11.60) | 115.64 (11.49) | 112.92 (15.52) | 86.87 (11.33) | 137.77 (11.50)
Statistical Analysis 1: Comparison: Placebo vs HB/APAP; Test type: Superiority; p = 0.3706, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs VX-548: Low Dose; Test type: Superiority; p = 0.5379, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs VX-548: Mid Dose; Test type: Superiority; p = 0.3859, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs VX-548: High Dose; Test type: Superiority; p = 0.0251, ANCOVA

2. Secondary Outcome: Time-Weighted SPID as Recorded on a NPRS 0 to 24 Hours (SPID24) After the First Dose of Study Drug
Description: SPID was calculated as the sum of the product of time (in hours) elapsed since previous measurements and pain intensity difference. Pain intensity difference was calculated by subtracting the pain intensity score at given post-dose time points from the baseline pain intensity scores (using pain rating score range: 0= no pain to 10= worst possible pain). SPID24 was calculated from 0 to 24 hours and the score range was -240 (worst score) to 240 (best score).
Time Frame: 0 to 24 hours After First Dose of Study Drug
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- HB/APAP: Participants received HB 5 mg/ APAP 325 mg capsule q6h for 2 days.
Arm/Group | Placebo | HB/APAP | VX-548: Low Dose | VX-548: Mid Dose | VX-548: High Dose
Number analyzed (Participants) | 59 | 60 | 33 | 62 | 60
units on a scale | 31.54 (5.57) | 40.95 (5.52) | 34.36 (7.45) | 24.78 (5.44) | 45.22 (5.52)
Statistical Analysis 1: Comparison: Placebo vs HB/APAP; Test type: Superiority; p = 0.2318, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs VX-548: Low Dose; Test type: Superiority; p = 0.7615, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs VX-548: Mid Dose; Test type: Superiority; p = 0.3870, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs VX-548: High Dose; Test type: Superiority; p = 0.0823, ANCOVA

3. Secondary Outcome: Percentage of Participants With at Least 30 Percent (%) Reduction in NPRS at 48 Hours After the First Dose of Study Drug
Description: Pain intensity was recorded on 11-point NPRS, score range: 0 to 10, where 0= no pain and 10= worst imaginable pain. The percentage of participants with at least 30% reduction from baseline in NPRS at 48 hours after the first dose of VX-548, HB/APAP or placebo was reported.
Time Frame: From Baseline at 48 Hours After First Dose of Study Drug
Population: FAS.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants received placebo and HB/APAP for 2 days.
Arm/Group | Placebo | HB/APAP | VX-548: Low Dose | VX-548: Mid Dose | VX-548: High Dose
Number analyzed (Participants) | 59 | 60 | 33 | 62 | 60
percentage of participants | 67.8 | 68.3 | 75.8 | 62.9 | 83.3
Statistical Analysis 1: Comparison: Placebo vs HB/APAP; Test type: Superiority; p = 0.9986, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs VX-548: Low Dose; Test type: Superiority; p = 0.4446, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs VX-548: Mid Dose; Test type: Superiority; p = 0.5978, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs VX-548: High Dose; Test type: Superiority; p = 0.0479, Cochran-Mantel-Haenszel

4. Secondary Outcome: Percentage of Participants With at Least 50% Reduction in NPRS at 48 Hours After the First Dose of Study Drug
Description: Pain intensity was recorded on 11-point NPRS, score range: 0 to 10, where 0= no pain and 10= worst imaginable pain. The percentage of participants with at least 50% reduction from baseline in NPRS at 48 hours after the first dose of VX-548, HB/APAP or placebo were reported.
Time Frame: From Baseline at 48 Hours After First Dose of Study Drug
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | HB/APAP | VX-548: Low Dose | VX-548: Mid Dose | VX-548: High Dose
Number analyzed (Participants) | 59 | 60 | 33 | 62 | 60
percentage of participants | 61.0 | 61.7 | 72.7 | 56.5 | 66.7
Statistical Analysis 1: Comparison: Placebo vs HB/APAP; Test type: Superiority; p = 0.9895, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs VX-548: Low Dose; Test type: Superiority; p = 0.2731, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs VX-548: Mid Dose; Test type: Superiority; p = 0.6492, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs VX-548: High Dose; Test type: Superiority; p = 0.5119, Cochran-Mantel-Haenszel

5. Secondary Outcome: Percentage of Participants With at Least 70% Reduction in NPRS at 48 Hours After the First Dose of Study Drug
Description: Pain intensity was recorded on 11-point NPRS, score range: 0 to 10, where 0= no pain and 10= worst imaginable pain. The percentage of participants with at least 70% reduction from baseline in NPRS at 48 hours after the first dose of VX-548, HB/APAP or placebo were reported.
Time Frame: From Baseline at 48 Hours After First Dose of Study Drug
Population: FAS.
Measure: Number; unit: percentage of participants
Groups:
- HB/APAP: Participants received HB 5 mg/ APAP 325 mg q6h 2 days.
Arm/Group | Placebo | HB/APAP | VX-548: Low Dose | VX-548: Mid Dose | VX-548: High Dose
Number analyzed (Participants) | 59 | 60 | 33 | 62 | 60
percentage of participants | 40.7 | 50.0 | 51.5 | 38.7 | 51.7
Statistical Analysis 1: Comparison: Placebo vs HB/APAP; Test type: Superiority; p = 0.3158, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs VX-548: Low Dose; Test type: Superiority; p = 0.3247, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs VX-548: Mid Dose; Test type: Superiority; p = 0.8424, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs VX-548: High Dose; Test type: Superiority; p = 0.2312, Cochran-Mantel-Haenszel

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of VX-548 and M6-548 (Metabolite)
Time Frame: Day 1 and Day 2
Population: Pharmacokinetic (PK) analysis set included participants who received at least 1 dose of VX-548. Here, "Number Analyzed" signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (mcg/mL)
Arm/Group | VX-548: Low Dose | VX-548: Mid Dose | VX-548: High Dose
Number analyzed (Participants) | 33 | 62 | 60
micrograms/milliliter (mcg/mL)
  VX-548: Day 1: number analyzed (Participants) | 31 | 58 | 58
  VX-548: Day 1 | 0.119 (0.0536) | 0.311 (0.0864) | 0.523 (0.193)
  VX-548: Day 2: number analyzed (Participants) | 29 | 55 | 57
  VX-548: Day 2 | 0.118 (0.0426) | 0.337 (0.0951) | 0.503 (0.126)
  M6-548: Day 1: number analyzed (Participants) | 31 | 58 | 58
  M6-548: Day 1 | 0.0929 (0.0363) | 0.234 (0.0781) | 0.385 (0.114)
  M6-548: Day 2: number analyzed (Participants) | 29 | 55 | 57
  M6-548: Day 2 | 0.183 (0.0520) | 0.483 (0.130) | 0.787 (0.210)

7. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of VX-548 and M6-548 (Metabolite)
Time Frame: Day 1 and Day 2
Population: PK analysis set included participants who received at least 1 dose of VX-548. Here, "Number Analyzed" signifies those participants who were evaluable at specified time points.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | VX-548: Low Dose | VX-548: Mid Dose | VX-548: High Dose
Number analyzed (Participants) | 33 | 62 | 60
hours (h)
  VX-548: Day 1: number analyzed (Participants) | 31 | 58 | 58
  VX-548: Day 1 | 2.20 [0.967 to 6.00] | 2.17 [1.00 to 5.98] | 2.09 [1.00 to 6.03]
  VX-548: Day 2: number analyzed (Participants) | 29 | 55 | 57
  VX-548: Day 2 | 1.93 [0.867 to 7.87] | 1.97 [0.850 to 6.00] | 2.00 [0.667 to 5.98]
  M6-548: Day 1: number analyzed (Participants) | 31 | 58 | 58
  M6-548: Day 1 | 6.00 [1.08 to 12.0] | 5.95 [2.00 to 12.2] | 6.02 [1.92 to 12.1]
  M6-548: Day 2: number analyzed (Participants) | 29 | 55 | 57
  M6-548: Day 2 | 5.88 [1.00 to 8.05] | 4.28 [1.00 to 12.0] | 4.20 [1.70 to 12.0]

8. Secondary Outcome: Area Under the Concentration Versus Time Curve From 0 to 12 Hours (AUC0-12h) of VX-548 and M6-548 (Metabolite)
Time Frame: Day 1 and Day 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hour*mcg/ml (h*mcg/mL)
Arm/Group | VX-548: Low Dose | VX-548: Mid Dose | VX-548: High Dose
Number analyzed (Participants) | 33 | 62 | 60
hour*mcg/ml (h*mcg/mL)
  VX-548: Day 1: number analyzed (Participants) | 29 | 51 | 57
  VX-548: Day 1 | 0.650 (0.173) | 1.84 (0.451) | 2.95 (0.745)
  VX-548: Day 2: number analyzed (Participants) | 28 | 55 | 57
  VX-548: Day 2 | 0.885 (0.248) | 2.54 (0.731) | 3.72 (0.873)
  M6-548: Day 1: number analyzed (Participants) | 29 | 51 | 57
  M6-548: Day 1 | 0.845 (0.337) | 2.23 (0.753) | 3.53 (1.13)
  M6-548: Day 2: number analyzed (Participants) | 27 | 52 | 56
  M6-548: Day 2 | 1.94 (0.577) | 5.12 (1.41) | 8.27 (2.16)

9. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Day 16
Population: Safety set included all participants who had received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- HB/APAP: Participants received HB/APAP 5 mg/ APAP 325 mg q6h for 2 days.
Arm/Group | Placebo | HB/APAP | VX-548: Low Dose | VX-548: Mid Dose | VX-548: High Dose
Number analyzed (Participants) | 59 | 60 | 33 | 62 | 60
Participants
  Participants with TEAEs | 23 | 25 | 7 | 17 | 18
  Participants with SAEs | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 16
Arm/Group | Placebo | HB/APAP | VX-548: Low Dose | VX-548: Mid Dose | VX-548: High Dose
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/60 | 0/33 | 0/62 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/60 | 0/33 | 0/62 | 0/60
Other Adverse Events (participants affected / at risk) | 12/59 | 13/60 | 2/33 | 7/62 | 9/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=59) | HB/APAP (N=60) | VX-548: Low Dose (N=33) | VX-548: Mid Dose (N=62) | VX-548: High Dose (N=60)
Nausea (Gastrointestinal disorders) | 5 | 11 | 2 | 3 | 5
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 0
Headache (Nervous system disorders) | 7 | 4 | 0 | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT04977336/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT04977336/SAP_001.pdf